CLINICAL TRIAL: NCT02743403
Title: Effects of Transcutaneous Electric Nerve Stimulation in Pain During Application of Carboxytherapy in Patients With Gynoid Lipodystrophy: Randomized Controlled Trial
Brief Title: Effects of TENS in Pain During Application of Carboxytherapy in Patients With Gynoid Lipodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Adria Yared Sadala, Clinical Researcher, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Carboxytherapy,TENS and pain
Record Dates: First submitted 2016-03-28; First posted 2016-04-19 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Neurodyn Portable TENS (Active Comparator): Subjects in this study arm will receive active treatment. The active TENS device will be Neurodyn Portable TENS the IBRAMED® and application of carboxytherapy device will be Carboxyderm S20-1C equipment, Tone Derm® brand.
  The subject receives both devices at the same time. The parameters of the active TENS are: frequency (f) of 100 Hertz (Hz) oscillator every 0.5 seconds pulse duration (T) 200 microseconds (microsiemens) and the amplitude (I) will be adjusted at the time of application the carboxiterapia.
  The application of Carboxytherapy is realized by a carboxy Derm S20-1C equipment Derm® mark, which uses carbon dioxide (CO2) medical and non-toxic.
  Each prick with a needle carboxiterapia will 100ml / min and will last 1 minute long.
  Before each puncture will be adjusted to the intensity of TENS as sensitivity of the subject.
  Interventions: Device: Neurodyn Portable activeTENS, IBRAMED®; Device: Neurodyn Portable placeboTENS, IBRAMED®; Device: Carboxyderm S20-1C
- Placebo TENS- Neurodyn Portable TENS (Placebo Comparator): Subjects in this study arm will receive placebo treatment. The placebo TENS device will be Neurodyn Portable TENS the IBRAMED® and application of carboxytherapy device will be Carboxyderm S20-1C equipment, Tone Derm® brand.
  The application of placebo TENS will be made by the same unit of active TENS; however, it is used a device specially developed for this study. The device remains active only during the first 30 seconds of application. After this time, the current amplitude will gradually decrease over the next 15 seconds until it reaches zero, thereby interrupting the emission of electrical power to the remainder of the application time. The display of placebo TENS device shows a light on all the time of application, indicating the patient that the device is active.
  Interventions: Device: Neurodyn Portable activeTENS, IBRAMED®; Device: Neurodyn Portable placeboTENS, IBRAMED®; Device: Carboxyderm S20-1C
- Control (No Intervention): Subjects in this study arm only receive the application carboxiterapia through Carboxyderm S20-1C equipment, Tone Derm® brand.
  The group (active - control Carboxytherapy) will be submitted to the application of Carboxytherapy and off TENS.

INTERVENTIONS:
Device: Neurodyn Portable activeTENS, IBRAMED® — Randomization and secret Allocation active TENS (GI / n = 27)
  Other Names: Carboxyderm S20-1C
  Arms: Neurodyn Portable TENS; Placebo TENS- Neurodyn Portable TENS
Device: Neurodyn Portable placeboTENS, IBRAMED® — Randomization and secret Allocation placebo TENS (GII / n = 27)
  Other Names: Carboxyderm S20-1C
  Arms: Neurodyn Portable TENS; Placebo TENS- Neurodyn Portable TENS
Device: Carboxyderm S20-1C — Randomization and secret Allocation control group (CG / n = 27).
  Arms: Neurodyn Portable TENS; Placebo TENS- Neurodyn Portable TENS

SUMMARY:
The project aims to compare the use of carboxiterapia ( therapeutic administration of carbon dioxide) with the use of active TENS and placebo TENS using the VAS scale as a parameter. The therapy used was started in the 30s , with carbonated water baths, and , lately, is involved in the therapeutic arsenal of numerous diseases , Both for treatment of diseases when for aesthetic treatments , especially for the gynoid lipodystrophy. However, the therapy presents CO2 in clinical practice, limiting factors for its use , such as pain at the injection site , small bruises or welts due to several punctures and feeling of crepitus. To try to combat these " side effects " that can last up to 30 minutes, the TENS was used in order to determine whether the use of this electric current helps at improvement of discomfort.

DETAILED DESCRIPTION:
The assessment and intervention will be carried out only by the researcher, which has physical therapy training and expertise in dermato-functional physiotherapy with clinical experience in 11 years, as well as fulfilling all the prerequisites required for the management of carboxytherapy, according the judgment 293 of 16 June 2012 the Federal Council of Physical Therapy and Occupational Therapy (COFFITO). Patients will be submitted for assessment and intervention once.

Assessments should contain demographic information of the participants by asking questions such as age, marital status, education and contact, lifestyle, gynecological history, surgical history, anthropometric measurements and physical inspection examination (Annex 3). Patients are advised not to make use of any medication for pain relief such as painkillers and anti-inflammatories, within 4 hours before the physiotherapy session. For physical examination, evaluations will be conducted in the standing position, with bathing suit, keeping the gluteal region with maximum visibility. The appraiser will inspect the bilateral gluteal region, to confirm the moderate degree of severity of the gynoid lipodystrophy, defined by the gynoid lipodystrophy severity scale, with the number of skin depressions (ND) in moderate amount, ND≥ 5-9 depressions, according CSS classification.

For the study, three groups will be divided: group A (active TENS + active Carboxytherapy), Y group (TENS placebo + active Carboxytherapy) and S (active - control Carboxytherapy). Group A (active TENS + active Carboxytherapy) will be submitted to the application of TENS during the application of Carboxytherapy, both linked. The Y group (TENS placebo + active Carboxytherapy) will be submitted to the application of Carboxytherapy and TENS with low-dose therapy. The group S (active - control Carboxytherapy) will be submitted to the application of Carboxytherapy and off TENS. Prior to the beginning of the study, both devices will be calibrated. The gluteal that receive the intervention will be defined by lot.

After drawing the group and laterality of the gluteal region that receive the intervention, will be marked by white pencil, the depressions of the skin with cellulite and the delimitation of the area, from the following lines: lateral line will have as midpoint the greater trochanter, where a vertical line will be drawn from the iliac crest to the lateral edge of the gluteal groove; top line will be drawn a horizontal line parallel to the gluteal groove, 4 cm below the posterior superior iliac spine to the vertical line drawn previously from the greater trochanter bottom line will be drawn a horizontal line delimiting the gluteal groove; the medial end of the gluteal groove to the vertical line drawn previously from the greater trochanter; medial line is delimited by anatomically intergluteal slot.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index < 18,5 a 29,9 kg/m²
* with regular menstrual cycle
* without prior experience with carboxytherapy and TENS
* with the presence of moderate gynoid lipodystrophy at gluteal region as classification Hexsel Dal'Forno & Hexsel (CSS )

Exclusion Criteria:

* pregnant women;
* nursing mothers;
* women with metabolic disorders and autoimmune diseases;
* which are suffering from skin lesions in the gluteal region and who have undergone surgical procedures in gluteus;
* the presence of malignant or benign tumor;
* with metal or silicone implants;
* heart disease and / or use of pacemakers, hypoesthesia or anesthesia in the gluteal region;
* women who have the risk of presenting epilepsy.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mesure and denouement | through study completion, an average of 1 year
  It will be used to assess pain intensity of the participants. This scale has 11 points, ranging from 0 to 10, where 0 is "no pain" and 10 "worst pain imaginable". Pain intensity will be measured in three groups: Group A, Group B and Group C, where the patient will quantify their pain viewing a rule containing a scale of 0 to 10. The assessment of this parameter will be made verbally, in which the patient should report the intensity of your pain when you are getting each prick of carboxytherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, PhD, Study Director
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes